CLINICAL TRIAL: NCT00305227
Title: Intravaginal LACTIN-V for Prevention of Recurrent Urinary Tract Infections
Brief Title: Intravaginal LACTIN-V for Prevention of Recurrent Urinary Tract Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Osel, Inc. (Industry)
Responsible Party: Principal Investigator, Ann Stapleton, Professor, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 28552; 5P01DK053369 (NIH); UW/LB-001 (Other: University of Washington)
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Urinary Tract Infection
Keywords: urinary tract infection; cystitis; Lactobacillus; probiotic; prevention
MeSH Terms: conditions — Urinary Tract Infections; Cystitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactin-V (Experimental): Vaginal capsule containing Lactobacillus crispatus in high concentration. Self-administered once daily for 5 days during the 1st week. Self-administered once weekly for 10 weeks.
  Interventions: Drug: Lactin-V
- Placebo (Placebo Comparator): Vaginal capsule - placebo. Self-administered once daily for 5 days during the 1st week. Self-administered once weekly for 10 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactin-V
  Other Names: no other names
  Arms: Lactin-V
Drug: Placebo
  Other Names: no other names
  Arms: Placebo

SUMMARY:
Recurrent urinary tract infections (RUTIS) continue to be a major health problem in women and are now complicated by increasing antibiotic resistance. New preventive approaches are needed. Because most women with RUTI lack the normal protective Lactobacillus (LB) in their vaginal flora, we hypothesized that restoration of LB would reduce RUTIS. In this trail, women with recent UTI are randomized to receive either LB or placebo vaginal capsules and are followed for side effects, for colonization with LB and for occurrence of RUTI over hte next four months.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to evaluate the safety of the vaginal suppository LACTIN-V (Lactobacillus crispatus CTV-05) as well as the efficacy of LACTIN-V use in preventing recurrent urinary tract infections (RUTI) in women. Study subjects will include pre-menopausal women with a history of frequent RUTI. As part of this study, we will also evaluate growth of lactobacilli and urinary tract infection(UTI)-causing bacteria in the vaginas of women following use of LACTIN-V.

Rationale: LACTIN-V is composed of L. crispatus. L. crispatus is a bacteria found to grow naturally in the vaginas of healthy women. It is felt to be important in preventing vaginal infection and UTI. With regard to prevention of UTI, L. crispatus is thought to prevent the growth of UTI-causing bacteria (such as E. coli) in the vagina, and so prevent these UTI-causing bacteria from being able to enter the female urethra and cause infection in the bladder (cystitis). There is epidemiologic evidence to support this prevention mechanism, as absence of L. crispatus and related lactobacilli from the vagina has been associated with vaginal E. coli growth and with UTI. Scientific evidence supports the ability of lactobacilli to prevent vaginal E. coli growth by out-competing E. coli in vaginal colonization, and through the production of toxins such as lactic acid, hydrogen peroxide, and bacteriocins.

LACTIN-V contains a specific strain of L. crispatus, CTV-05, which was isolated from the vagina of a healthy woman. It was prepared as a vaginal suppository with the purpose of restoring growth of healthy L. crispatus in the vaginas of women who experience frequent RUTI. As indicated above, these women often have a deficiency of healthy vaginal lactobacilli growth, and therefore may not experience the protective function of these natural organisms. It is hoped that use of LACTIN-V will lead to vaginal growth of protective lactobacilli in these women wich will, in turn, prevent the vaginal growth of E. coli and other UTI-causing bacteria. Phase 1 and 2 studies of LACTIN-V to date have shown this "probiotic" to be safe and well tolerated.

The impetus for this study is the urgent need for non-antibiotic strategies to prevent UTI. UTI is one of the most common bacterial infections. It leads to substantial morbidity and health care costs. Frequent use of antibiotics for treatment of and prophylaxis against UTI is contributing to the prevalence of antibiotic resistant bacteria, which are also making it more difficult to treat UTI. Therefore, the potential advantage of LACTIN-V is that it is a natural product that may prevent UTI without the use of antibiotics. If it proves to be efficacious, it could decrease the morbidity and health care costs associated with UTI as well as decrease overall antibiotic use and the corresponding prevalence of antibiotic resistance among UTI-causing bacteria.

Primary Objective: The primary objective is to evaluate the safety of LACTIN-V, compared to placebo, in pre-menopausal women with recurrent uncomplicated UTI.

Secondary objectives:

1. To evaluate the efficacy of LACTIN-V, compared to placebo, in reducing the incidence of Symptomatic and Probable UTI (defined below).
2. To evaluate the efficacy of LACTIN-V, compared to placebo, in decreasing the time to recurrence of Symptomatic and Probable UTI.
3. To evaluate the efficacy of LACTIN-V, compared to placebo, in reducing the prevalence of Asymptomatic UTI (defined below).
4. To evaluate vaginal growth of CTV-05 in subjects using LACTIN-V compared to placebo.
5. To evaluate vaginal growth of lactobacilli in subjects using LACTIN-V compared to subjects using placebo.
6. To evaluate vaginal growth of E. coli in subjects using LACTIN-V compared to subjects using placebo.

Case Definitions:

Symptomatic UTI: One or more UTI symptoms (dysuria, urgency, frequency, suprapubic pain, flank pain), with a positive urine culture. In symptomatic subjects, a positive urine culture is defined as >= 10^2/ml of an UTI-causing bacteria. UTI episodes will be recorded as Symptomatic UTI if a negative urine culture at Visit 2, or at another interim study visit, confirms resolution of the prior UTI (in order to distinguish a new Symptomatic UTI from a Persistent UTI).

Asymptomatic UTI: A positive urine culture in a subject who reports no urinary symptoms. In asymptomatic subjects, a positive urine culture is defined as >= 10^5/ml of an UTI-causing bacteria. UTI episodes will be recorded as Asymptomatic UTI if a negative urine culture at Visit 2, or at another interim study visit, confirms resolution of the prior UTI (in order to distinguish a new Asymptomatic UTI from a Persistent UTI).

Probable UTI: One or more UTI symptoms (dysuria, urgency, frequency, suprapubic pain, flank pain) in a subject who contacted a healthcare provider and was treated with antibiotics for a UTI without confirmatory urine culture. UTI episodes will be recorded as Probable UTI if a negative urine culture at Visit 2, or at another interim study visit, confirms resolution of the prior UTI (in order to distinguish a new Probable UTI from a Persistent UTI).

Persistent UTI: A positive urine culture following antibiotic treatment for a UTI.

General Procedures: This will be a randomized, double-blind, placebo-controlled trial of LACTIN-V. Subjects will include 100 pre-menopausal women with a history of frequent RUTI who are currently or recently being treated for a symptomatic UTI with trimethoprim-sulfamethoxazole. Trimethoprim-sulfamethoxazole is one of several antibiotics considered standard-of-care for treatment of symptomatic UTI. Subjects will be randomized such that 50 women will receive LACTIN-V at a dose of 5x10^8 CFU/suppository and 50 women will receive placebo. LACTIN-V and placebo are to be taken once per day for five days during the first week of use followed by once per week for 10 weeks on Days 8, 15, 22, 29, 36, 43, 50, 57, 64, and 71 for a total of 15 doses over 11 weeks. Subjects will undergo five scheduled visits and receive two telephone calls:

Visit 1 is the Screening Visit. This visit will take place during or soon after evaluation for a symptomatic UTI. The following will occur during Visit 1: informed consent, review of eligibility, history, physical exam, pelvic exam, Pap smear, urine pregnancy test, and screening tests for gonorrhea, chlamydia, bacterial vaginosis, yeast, and trichomonas. Subjects will provide urine samples for microscopic analysis, dipstick analysis, culture, and antibiotic susceptibility testing and vaginal fluid specimens for laboratory assessment of vaginal growth of lactobacilli (including CTV-05).

Visit 2 is the Randomization Visit and represents Week 1 of the study. Visit 2 will take place 3-10 days after completion of antibiotic therapy for UTI. Subjects will have their eligibility confirmed and undergo a focused pelvic exam without speculum or bimanual exam unless clinically indicated, have a screening test for bacterial vaginosis, yeast, and trichomonas, and have a repeat pregnancy test. Subjects will also provide urine and vaginal fluid specimens as in Visit 1. Subjects will then be randomized to LACTIN-V or placebo. Subjects will place the first suppository under supervision and will be instructed to use a 7-day study calendar to record study product use and related symptoms during the first week, and to use a 10-week study calendar to record study product use and related symptoms thereafter.

Day 4-7 phone call: The purpose of this phone call is to assess use of the study product as well as any associated symptoms.

Visit 3 will occur during Week 2, days 8-14 following randomization. Subjects will be asked about study product use, adverse events, and symptoms. Subjects will undergo focused physical and pelvic exams without speculum or bimanual exam unless clinically indicated. Subjects will have a screening test for bacterial vaginosis and provide urine and vaginal fluid specimens as before.

Visit 4 will occur during Week 11 and will be similar to Visit 3.

Visit 5 will occur during Week 16. The procedures for Visit 5 will be similar to those of Visits 3 and 4. However, during this visit, subjects will undergo a complete pelvic exam including speculum and bimanual exams and undergo a repeat pregnancy test.

9 Month telephone call: The purpose of this phone call is to assess the occurrence of adverse events, symptoms of UTI, new UTI or other medical diagnoses,and pregnancy.

In addition to the above schedules visits, subjects will be asked to come to the research clinic for Unscheduled Visits if they experience any adverse events or new symptoms of UTI. During these unscheduled visits, subjects will undergo history, physical and complete pelvic exams, screening tests for bacterial vaginosis, yeast, and trichomonas, as well as for other sexually transmitted diseases as clinically indicated. Subjects will provide urine samples for microscopic analysis, dipstick analysis, culture, and antibiotic susceptibility testing. Subjects will provide vaginal fluid samples for assessment of CTV-05, lactobacillus, and E. coli growth.

Subjects diagnosed with a Symptomatic UTI during the study will be treated with an antibiotic. They will then be asked to return to the study clinic for a follow-up urine culture two weeks later to confirm UTI resolution.

Laboratory procedures will include:

* wet mount slides of vaginal fluid (all Visits)
* urine dipstick testing (all Visits)
* urine pregnancy testing (Visits 1, 2, and 5)
* Pap smear (Visit 1)
* Testing for gonorrhea and chlamydia by culture (Visit 1, other visits as indicated)
* urinalysis (all Visits)
* urine culture (all Visits)
* gram stain and culture of vaginal fluid specimens (All Visits)
* Rep-PCR for CTV-05 (Visits 2-5)
* DNA amplification of vaginal flora (all Visits)

Statistical Analysis: The primary cohort for analysis will be the intent-to-treat (ITT) cohort. The ITT cohort is defined as subjects who are randomized in the study. Other cohorts to be evaluated will include the modified ITT, Evaluable, and according-to-protocol cohorts.

ELIGIBILITY:
Inclusion Criteria:

* pre-menopausal woman aged 18-40 years
* current symptomatic uncomplicated cystitis
* cystitis is treated with trimethoprim-sulfamethoxazole (TMP-SMX)
* completion of screening procedures
* negative screening monolayer Pap smear or hysterectomy
* history of at least two prior symptomatic UTI's treated within the past 12 months or one pior symptomatic UTI treated in the past six months
* agree to return for the Randomization Visit (Visit 2)
* regular menstrual cycles or amenorrheic due to use of a long acting progestin, continuous use of oral contraceptives or hysterectomy
* willing to insert vaginal capsules without an applicator
* capable of providing informed consent
* able to read and understand English
* agree to abstain from self-medication with antibiotics for UTI symptoms
* agree to abstain from antibiotic prophylaxis for recurrent UTI
* agree to abstain from the use of any other intra-vaginal product
* agree to abstain from sexual intercourse for 24 hours after capsule insertion
* agree to not use tampons for 24 hours after capsule insertion
* agree to use an adequate method of birth control

Exclusion Criteria:

* complicated cystitis or uncomplicated pyelonephritis.
* cystitis at Visit 1 not treated with TMP-SMX
* uropathogen resistant to TMP-SMX isolated at Visit 1 and persistent symptoms at Visit 2 or failure to achieve a significant reduction in urine wbc count at Visit 2
* vaginal or cervical infection, currently or within the past 21 days, with bacterial vaginosis (treated, symptomatic infection), Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis or Herpes Simplex
* symptomatic bacterial vaginosis at Visit 1
* high risk for sexually transmitted diseases and/or HIV, including:

  1. diagnosis of N. gonorrhoeae, C. trachomatis or T. vaginalis on two or more occasions during the previous six months;
  2. sexual intercourse with a homosexual/bisexual male in the last 10 years;
  3. sexual intercourse with an injection drug user or sex worker in the last 10 years; or
  4. shared needles for injected drugs in the last 10 years.
* chronic vaginal, urinary or pelvic symptoms not attributable to UTI
* recurrent bacterial vaginosis (three or more symptomatic, treated infections in the prior 12 months)
* pregnancy or within two months of last pregnancy
* lactation
* antibiotic therapy fewer than three days prior to Randomization Visit
* antifungal therapy fewer than seven days prior to the Randomization Visit
* Antibiotics planned within four months
* abnormal Pap smear requiring a procedure for diagnosis or treatment in the past 12 months
* use of CTV-05 within one year of the Randomization Visit
* menopause
* use of a NuvaRing planned during the course of the study
* any significant disease or acute illness that in the Investigator's assessment could complicate the evaluation
* known HIV infection
* immunosuppressive drug within 60 days
* known allergy to any component of LACTIN-V or the placebo capsule
* unavailable for follow-up visits
* drug or alcohol abuse within past two years
* any social or medical condition that, in the opinion of the Investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2006-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann E Stapleton, MD, Principal Investigator — University of Washington
Locations (1):
- Hall Health Primary Care Center, University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Giorgi A, Torriani S, Dellaglio F, Bo G, Stola E, Bernuzzi L. Identification of vaginal lactobacilli from asymptomatic women. Microbiologica. 1987 Oct;10(4):377-84. PMID 3695985
- [Background] Antonio MA, Hawes SE, Hillier SL. The identification of vaginal Lactobacillus species and the demographic and microbiologic characteristics of women colonized by these species. J Infect Dis. 1999 Dec;180(6):1950-6. doi: 10.1086/315109. PMID 10558952
- [Background] Antonio MA, Hillier SL. DNA fingerprinting of Lactobacillus crispatus strain CTV-05 by repetitive element sequence-based PCR analysis in a pilot study of vaginal colonization. J Clin Microbiol. 2003 May;41(5):1881-7. doi: 10.1128/JCM.41.5.1881-1887.2003. PMID 12734221
- [Background] Foxman B, Barlow R, D'Arcy H, Gillespie B, Sobel JD. Urinary tract infection: self-reported incidence and associated costs. Ann Epidemiol. 2000 Nov;10(8):509-15. doi: 10.1016/s1047-2797(00)00072-7. PMID 11118930
- [Background] Stamm WE, Counts GW, Wagner KF, Martin D, Gregory D, McKevitt M, Turck M, Holmes KK. Antimicrobial prophylaxis of recurrent urinary tract infections: a double-blind, placebo-controlled trial. Ann Intern Med. 1980 Jun;92(6):770-5. doi: 10.7326/0003-4819-92-6-770. PMID 6992677
- [Background] Gupta K, Scholes D, Stamm WE. Increasing prevalence of antimicrobial resistance among uropathogens causing acute uncomplicated cystitis in women. JAMA. 1999 Feb 24;281(8):736-8. doi: 10.1001/jama.281.8.736. PMID 10052444
- [Background] Hooton TM, Scholes D, Gupta K, Stapleton AE, Roberts PL, Stamm WE. Amoxicillin-clavulanate vs ciprofloxacin for the treatment of uncomplicated cystitis in women: a randomized trial. JAMA. 2005 Feb 23;293(8):949-55. doi: 10.1001/jama.293.8.949. PMID 15728165
- [Background] Reid G, Bruce AW, Fraser N, Heinemann C, Owen J, Henning B. Oral probiotics can resolve urogenital infections. FEMS Immunol Med Microbiol. 2001 Feb;30(1):49-52. doi: 10.1111/j.1574-695X.2001.tb01549.x. PMID 11172991
- [Background] Stamey TA, Sexton CC. The role of vaginal colonization with enterobacteriaceae in recurrent urinary infections. J Urol. 1975 Feb;113(2):214-7. doi: 10.1016/s0022-5347(17)59447-1. PMID 803573
- [Background] Gupta K, Stapleton AE, Hooton TM, Roberts PL, Fennell CL, Stamm WE. Inverse association of H2O2-producing lactobacilli and vaginal Escherichia coli colonization in women with recurrent urinary tract infections. J Infect Dis. 1998 Aug;178(2):446-50. doi: 10.1086/515635. PMID 9697725
- [Background] Hooton TM, Fihn SD, Johnson C, Roberts PL, Stamm WE. Association between bacterial vaginosis and acute cystitis in women using diaphragms. Arch Intern Med. 1989 Sep;149(9):1932-6. PMID 2673116
- [Background] Hooton TM, Roberts PL, Stamm WE. Effects of recent sexual activity and use of a diaphragm on the vaginal microflora. Clin Infect Dis. 1994 Aug;19(2):274-8. doi: 10.1093/clinids/19.2.274. PMID 7986899
- [Background] Osset J, Bartolome RM, Garcia E, Andreu A. Assessment of the capacity of Lactobacillus to inhibit the growth of uropathogens and block their adhesion to vaginal epithelial cells. J Infect Dis. 2001 Feb 1;183(3):485-91. doi: 10.1086/318070. Epub 2000 Dec 29. PMID 11133381
- [Derived] Stapleton AE, Au-Yeung M, Hooton TM, Fredricks DN, Roberts PL, Czaja CA, Yarova-Yarovaya Y, Fiedler T, Cox M, Stamm WE. Randomized, placebo-controlled phase 2 trial of a Lactobacillus crispatus probiotic given intravaginally for prevention of recurrent urinary tract infection. Clin Infect Dis. 2011 May;52(10):1212-7. doi: 10.1093/cid/cir183. Epub 2011 Apr 14. PMID 21498386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 2006 ~ February 2009 University of Washington student health center
Period: Overall Study
Arm/Group | Lactin-V | Placebo
Started | 50 | 50
Completed | 43 (with at least 8 weeks of observation) | 44 (with at least 8 weeks of observation)
Not Completed | 7 | 6
Not completed — Lost to Follow-up | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactin-V | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 21 (18-31) [18 to 31] | 21 (18-36) [18 to 36] | 21 (18-36) [18 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Urinary Tract Infection
Description: Recurrent urinary tract infection after initiation of intervention. Culture-confirmed to contain uropathogen.
Time Frame: 10 weeks
Population: The reported analysis was by intention to treat. All study participants were used, except for 4 participants in whom the major outcome measure was unevaluable.
Measure: Number; unit: participants
Arm/Group | Lactin-V | Placebo
Number analyzed (Participants) | 48 | 48
participants | 7 | 13

2. Secondary Outcome: Incidence of Vaginal Discharge
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- Lactin-V: Vaginal capsule containing Lactobacillus crispatus in high concentration. Self-administered once daily for 5 days during the 1st week. Self-administered once weekly for 10 weeks.
  Lactin-V
- Placebo: Vaginal capsule - placebo. Self-administered once daily for 5 days during the 1st week. Self-administered once weekly for 10 weeks.
  Placebo
Arm/Group | Lactin-V | Placebo
Number analyzed (Participants) | 50 | 50
Participants | 4 | 5

ADVERSE EVENTS:
Time Frame: 10 weeks for serious adverse events
Description: Other adverse events (minor side effects) information was collected after the first week of intense(5 doses) dosing. The results presented were not specifically elicited by type of effect, i.e. they were not prompted for the nature of their side effect.
Arm/Group | Lactin-V | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 28/50 | 25/50
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lactin-V (N=50) | Placebo (N=50)
Painful urination (Renal and urinary disorders) | 1 | 2
Urinary frequency (Renal and urinary disorders) | 0 | 1
Pain in lower abdomen (General disorders) | 0 | 1
Low back pain (General disorders) | 0 | 1
Other urinary symptoms (Renal and urinary disorders) | 2 | 0
Vaginal odor (Reproductive system and breast disorders) | 3 | 4
Abnormal vaginal discharge (Reproductive system and breast disorders) | 4 | 5
Vaginal itch (Reproductive system and breast disorders) | 5 | 3
Painful intercourse (General disorders) | 1 | 0
Redness/irritation of genitals (General disorders) | 2 | 0
Genital swelling (General disorders) | 2 | 0
Other vaginal symptoms (Reproductive system and breast disorders) | 20 | 17
Diarrhea (General disorders) | 1 | 1
Abdominal discomfort (General disorders) | 1 | 1
Other symptoms (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No